CLINICAL TRIAL: NCT03272659
Title: The Correlation of Surgical Colorectal Cancer Specimen Pathology With the Fluorescence of Photodynamic Diagnostics (PDD): a Clinical Pilot Study
Brief Title: The Correlation of Surgical Colorectal Cancer Specimen Pathology With the Fluorescence of Photodynamic Diagnostics
Acronym: PDD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Long process and due to strict deadline, project was stopped.
Sponsor: Dr. Te Vuong (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Te Vuong, Director, Radiation Oncology Department, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-140
Record Dates: First submitted 2017-08-30; First posted 2017-09-05 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer; Photodynamic Diagnosis
Keywords: Fluorescence Sigmoidoscopy; PDD; Photodynamic Diagnosis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blue Light Cystoscopy with Cysview® (Experimental): The enema will be administered to participant. Fluorescence sigmoidoscopy will be performed with white light then blue excitation light after retention of the enema for 60 minutes, followed by a rest time of up to 30 minutes before rectoscopy.
  Post-operative surgical specimens will be collected for further fluorescence microscopy studies and pathological correlation of fluoresce with malignant pathology/histology as the gold standard.
  Interventions: Drug: Cysview

INTERVENTIONS:
Drug: Cysview — 250 mL enema containing 1.6 mmol of hexaminolevulinate
  Other Names: hexaminolevulinate

SUMMARY:
This will be a pilot study involving 5 patients diagnosed with colorectal carcinoma and treated with pre-operative chemotherapy and external beam radiation therapy at the Jewish General Hospital, whom will very soon undergo surgery. Participants will be sensitized by the instillation of a 250 mL enema containing 1.6 mmol of HAL. The enema will be administered with a plastic tube with an inflatable blocking balloon to prevent leakage of the enema. Fluorescence sigmoidoscopy will be performed with white light then blue excitation light after retention of the enema for 60 minutes, followed by a rest time of up to 30 minutes before rectoscopy. Red fluorescence should be induced by illumination with blue light. Pictures with and without fluorescence will be taken. The patients will undergo a colectomy (partial or complete) within the next 2-3 days and the surgical specimens will be collected for further fluorescence microscopy studies and pathological correlation of fluoresce with malignant pathology/histology as the gold standard. The total concentration of porphyrins in the patients' urine and serum will be recorded before sensitization, immediately after sensitization (instillation of the enema), and approximately 24 hours after sensitization. The patients' pre-and-post operative liver function tests will be measured. Adverse events will be reported by direct questioning of all patients with regards to photosensitivity and gastrointestinal symptoms (nausea, vomiting), and by measuring blood pressure and heart rate. Our objectives and endpoints are: 1) to determine if fluorescence with photodynamic diagnostics is selective for colorectal cancer, 2) to determine if photodynamic diagnostics has the potential to improve the detection of malignant cell after neoadjuvant chemotherapy and radiation, and 3) to determine if photodynamic diagnostics can provide an accurate depiction of the extent of disease burden not visible with normal white light sigmoidoscopy to the naked human eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age with diagnosed colorectal cancer.
* Colorectal cancer patients treated with Chemotherapy and external beam radiation therapy

Exclusion Criteria:

* 1) Liver cirrhosis
* 2) Acute or chronic hepatitis
* 3) Elevated liver function tests of unknown etiology with elevation of transaminases of more than 3 times normal levels
* 4) Known porphyria
* 5) Pregnancy
* 6) Expected lack of compliance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
fluorescence with photodynamic diagnostics (PDD) in colorectal cancer | 9 months
  To observe red fluorescence wirh PDD when lesions are illuminate with blue fluorescence during fluorescence sigmoidoscopy.

SECONDARY OUTCOMES:
Detect malignant lesions | 9 months
  Using the images of fluorescence sigmoidoscopy, detect malignant lesions after neoadjuvant chemotherapy and radiation.

OTHER OUTCOMES:
Accurate depiction of the extent of disease burden by correlating pre-and post surgical results after neoadjuvant chemotherapy and radiation. | 9 months

REFERENCES:
- [Background] Endlicher E, Gelbmann CM, Knuchel R, Furst A, Szeimies RM, Golder SK, Scholmerich J, Lottner C, Messmann H. Hexaminolevulinate-induced fluorescence endoscopy in patients with rectal adenoma and cancer: a pilot study. Gastrointest Endosc. 2004 Sep;60(3):449-54. doi: 10.1016/s0016-5107(04)01723-7. PMID 15332045
- [Background] Mayinger B, Neumann F, Kastner C, Degitz K, Hahn EG, Schwab D. Early detection of premalignant conditions in the colon by fluorescence endoscopy using local sensitization with hexaminolevulinate. Endoscopy. 2008 Feb;40(2):106-9. doi: 10.1055/s-2007-967019. Epub 2008 Jan 16. PMID 18197583
- [Background] Mayinger B, Neumann F, Kastner C, Haider T, Schwab D. Hexaminolevulinate-induced fluorescence colonoscopy versus white light endoscopy for diagnosis of neoplastic lesions in the colon. Endoscopy. 2010 Jan;42(1):28-33. doi: 10.1055/s-0029-1243804. Epub 2010 Jan 11. PMID 20066590
- [Background] Pietzak EJ. The Impact of Blue Light Cystoscopy on the Diagnosis and Treatment of Bladder Cancer. Curr Urol Rep. 2017 May;18(5):39. doi: 10.1007/s11934-017-0685-8. PMID 28324275
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787